CLINICAL TRIAL: NCT05680844
Title: Observational Study of the Correlation Between Peripheral Treg Cell Senescence and Serum Total Cholesterol Level
Brief Title: Peripheral Treg Cell Senescence & Serum Total Cholesterol Level
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xintong Ge, Professor, Tianjin Medical University General Hospital
Other Study IDs: IRB2022-YX-244-01
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hypercholesterolemia
Keywords: Treg; cell senescence; hypercholesterolemia; total cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal cholesterol level group: Serum total cholesterol level of < 5.17 mmol/L
- hypercholesterolemia group: Serum total cholesterol level of >= 5.17 mmol/L

SUMMARY:
Hypercholesterolemia is a risk factor for the occurrence and development of atherosclerosis. Recent animal studies have found that increased serum cholesterol level is associated with peripheral Treg cell senescence, but clinical evidence is still lacking. The purpose of this study is to analyze the correlation between human peripheral Treg cell senescence and serum total cholesterol level using clinical blood samples, thus laying a foundation for the establishment of novel therapeutic strategies for atherosclerosis based on the regulation of Treg cell senescence.

DETAILED DESCRIPTION:
Hypercholesterolemia is a risk factor for the occurrence and development of atherosclerosis. Recent animal studies have found that increased serum cholesterol level is associated with peripheral Treg cell senescence, but clinical evidence is still lacking. The purpose of this study is to analyze the correlation between human peripheral Treg cell senescence and serum total cholesterol level using clinical blood samples, thus laying a foundation for the establishment of novel therapeutic strategies for atherosclerosis based on the regulation of Treg cell senescence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 and ≤ 60 years old with independent behavior ability.
2. The participants need to fully understand the purpose and content of the study, and voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Acute and severe diseases in the last 3 months, including but not limited to, acute myocardial infarction, acute cerebral infarction, cerebral hemorrhage, circulatory failure, respiratory failure (internal diseases), trauma requiring hospitalization, or undergoes surgery under general anesthesia (surgical diseases).
3. History of severe diseases, including but not limited to, tumors, serious hematological diseases, serious cardiopulmonary diseases (interventional therapy for coronary artery disease, atrial fibrillation, chronic obstructive pulmonary disease, etc.), renal failure, liver failure, old stroke with serious sequelae.
4. Have participated in clinical trials in the past 3 months.
5. The investigator considers that not appropriate for inclusion.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 200 subjects were randomly selected from the population receiving physical examination in the Cadre Physical examination Center of Tianjin Medical University General Hospital from January 2023 to March 2023.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Treg cell senescence | After confirming the subject has signed the informed consent, and recorded the past medical history and medication (especially hypolipidemic drugs) in the past 3 months.
  Treg cell senescence will be evaluated by the beta-galactosidase (SA-betagal) activity test

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lei, Ph.D., Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05680844/Prot_000.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05680844/ICF_001.pdf